CLINICAL TRIAL: NCT01740232
Title: A Simple Trephination Increase the Heeling Potential for All-inside Meniscal Repair in the Vascular Zone
Brief Title: Can a Simple Trephination Increase the Heeling Potential for All-inside Meniscal Repair in the Vascular Zone?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mikkel Lindegaard Attrup (Other)
Responsible Party: Sponsor-Investigator, Mikkel Lindegaard Attrup, Staff Specialist 1, Amager Hospital
Organization: Amager Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: meniskprojekt; H-4-2012-093 (Other: Committee on Health Research Ethics)
Record Dates: First submitted 2012-10-12; First posted 2012-12-04 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Rupture; Meniscus, Bucket Handle
MeSH Terms: conditions — Rupture | interventions — Trephining

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trephination (Active Comparator): A 1 x 10 mm pricker are used for the trephination of the meniscus before normal meniscal repair.
  Interventions: Procedure: trephination
- Normal meniscal repair (Placebo Comparator): standard operation. Normal meniscalrepair.
  Interventions: Procedure: Normal meniscal repair

INTERVENTIONS:
Procedure: trephination — Artroscopic meniskal repair with trephination.
  Arms: Trephination
Procedure: Normal meniscal repair — Artroscopic meniskal repair without trephination.
  Other Names: Normal meniscal suture with FastFix device.
  Arms: Normal meniscal repair

SUMMARY:
Meniscus does not always heal when sutured. The investigators will make small holes in the meniscus before repair to promote more bleeding. The investigators expect that will help the meniscus to heal better.

DETAILED DESCRIPTION:
RCT study to evaluate the effect on trephination together with meniscal repair on meniscus healing after repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults who have a meniscus repaired.

Exclusion Criteria:

* Meniscus not fit for repair.
* Patients not fit for the repair regime.
* Arthrosis > stadie 2 (ICRS).
* Prior attempt of repair of the meniscus.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
KOOS Questionnaire | 4 month
  Primary outcome are differences between the to arms in the most relevant subgroup "Function, sports and recreational activities" in the KOOS questionnaire.
KOOS Questionnaire | 12 month
  Primary outcome are differences between the to arms in the most relevant subgroup "Function, sports and recreational activities" in the KOOS questionnaire.

SECONDARY OUTCOMES:
Clinical meniscus healing | 4 month

OTHER OUTCOMES:
Lysholm | 4 month
  Lysholm questionnaire
rearthroscopy | 6 month
KOOS | 12 month
  Differences between the to arms in the complete KOOS questionnaire.
Lysholm | 12 month
  Lysholm questionnaire
IKDC | 12 month
  IKDC questionnaire
IKDC | 4 month
  IKDC questionnaire
KOOS | 4 month
  Differences between the to arms in the complete KOOS questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Attrup, Principal Investigator — Artroscopic Center Amager
Locations (2):
- Denmark (2):
  - Artroskopisk Center Amager, Copenhagen S, Copenhagen
  - Artroskopisk Center Amager, Copenhagen